CLINICAL TRIAL: NCT00984581
Title: A Single-site, Double-blind Trial to Investigate the Safety, Tolerability, Systemic Exposure and Anti-scarring Potential of Intradermal Juvista in Female Subjects Aged 18-45 Years
Brief Title: Safety and Efficacy Study of Avotermin (Juvista) in Female Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Medical Director, Renovo Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RN1001-319-1006
Record Dates: First submitted 2009-09-15; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing
Keywords: Cicatrix; Scar; Wound healing; Avotermin; TGF beta 3; Juvista; RN1001
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Ltbp3 protein, zebrafish

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal avotermin (Experimental)
  Interventions: Drug: Avotermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avotermin — Intradermal injection, 5ng/100ul/linear cm wound margin administered on Day 0, Day 1 and month 6
  Other Names: TGFbeta 3; Juvista
  Arms: Intradermal avotermin
Drug: Avotermin — Intradermal injection, 50ng/100ul/linear cm wound margin administered on Day 0, Day 1 and month 6
  Other Names: TGFbeta 3; Juvista
  Arms: Intradermal avotermin
Drug: Placebo — Intradermal injection, 100ul/linear cm wound margin administered on Day 0 and Day 1
  Arms: Placebo

SUMMARY:
To assess safety and toleration, systemic exposure and anti-scarring potential of intradermal avotermin (Juvista) in young females.

DETAILED DESCRIPTION:
Subjects were to receive two 1cm incisions on the upper, inner aspect of each arm (four wounds per subject).

On Day 0 all subjects received intradermal Juvista at a concentration of 50ng/100ul to one incision site on Arm 1 and 5ng/100ul to one incision site on Arm 2. The other incision sites were injected with placebo. Following injection, 1cm incision wounds were made at each site.

On Day 1 all subjects were re-injected with 100ul/cm intradermal Juvista or placebo to each side of the wound (200ul per incision) at the same concentration as for Day 0 (50 or 5ng/100ul).

At month 6 all incision sites were excised for histological analysis and all excision sites injected with Juvista. Both sites on Arm 1 received 50ng/100ul/linear cm wound margin and both sites on Arm 2 received 5ng/100ul/linear cm wound margin. No excision sites received placebo.

The appearance of excision scars was then assessed after 2, 4 and 6 months of healing i.e at months 8, 10 and 12 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy, female subjects aged 18-45 years
* Weight between 40-150 kg and a BMI within the permitted range for their height using Quetelet's index (15-35 kg/m(squared)). Weight(kg)/height (squared)(m)
* Subjects who use appropriate non-pharmaceutical methods of contraception or are not likely to become pregnant for the duration of the trial

Exclusion Criteria:

* Subjects who have history or evidence of hypertrophic or keloid scarring or with tattoos or previous scars in the area to be biopsied
* Subjects with a personal history of a bleeding disorder
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring
* Subjects with a skin disorder that is chronic or currently active and which the investigator considers will adversely affect the healing of acute wounds or will involve the areas to be examined in this trial
* Subjects with any clinically significant medical condition that would impair wound healing including significant rheumatoid arthritis, chronic renal impairment, significant hepatic impairment, inadequately or uncontrolled digestive heart failure, active malignancy, immunosuppressive, radiation or chemotherapy within the last three months, a history of radiotherapy to the arm or diabetes mellitus
* Subjects with a history of clinically significant drug hypersensitivity to lignocaine or allergy to surgical dressings to be used in this trial
* Subjects with any clinically significant abnormality following review of pre-trial laboratory data and physical examination
* Subjects who are taking, or have taken, any investigational drugs, long term oral, topical or inhaled corticosteroid therapy, HRT, oral contraceptive pill, other pharmaceutical methods of contraception or anticoagulant drugs in the thirty days prior to Day 0
* Subjects who have evidence of drug abuse
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen or hepatitis C antibody. Subjects with previous vaccination against hepatitis B are not excluded per se
* Subjects who are carriers of the hepatitis B core antibody and who show less than 10 units per litre of Anti-HBs
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high risk group and subjects who at any point have a positive pregnancy test
* Subjects who are pregnant or become pregnant during the trial
* In the opinion of the investigator, a subject who is not likely to complete the trial for what ever reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2003-04; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To collect safety and tolerability data for intradermal injection of Juvista in a young female subject group. | Month 6

SECONDARY OUTCOMES:
To assess systemic exposure following intradermal Juvista before and after minor skin incisions. | Month 6
To assess the anti-scarring potential of intradermal Juvista in a young female population. | Month 6-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duncan, Principal Investigator — Renovo; Jeremy Bond, Principal Investigator — Renovo
Locations (1):
- Renovo, Manchester, United Kingdom